CLINICAL TRIAL: NCT05826106
Title: R Anastomosis for B-Ⅱ-B Anastomosis
Brief Title: The Benefits of R Anastomotic Technique for Billroth-Ⅱ Reconstruction With Braun Anastomosis After Totally Laparoscopic Distal Gastrectomy
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Jiajie Zhou, DR, Northern Jiangsu People's Hospital
Other Study IDs: NorthernJiangsuhospital
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Time for R Anastomosis; Complication Related to Anastomosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- R anastomosis
  Interventions: Procedure: R anastomosis

INTERVENTIONS:
Procedure: R anastomosis — Modifying the surgical technique of totally laparoscopic Billroth-II reconstruction with Braun anastomosis and to name it as the R anastomosis.

SUMMARY:
This study proposes a novel, straightforward, and viable technique for performing posterior gastrojejunostomy anastomosis during totally laparoscopic Billroth-II reconstruction with Braun anastomosis (named R anastomosis). This study prospectively evaluated clinical and pathological data from patients who underwent totally laparoscopic distal gastrectomy with R anastomosis at Northern Jiangsu People's Hospital, China, in order to investigate the feasibility and functional outcomes of R anastomosis for B-II-B anastomosis.

DETAILED DESCRIPTION:
Paients were recruited who were confirmed to have malignant tumors in the gastric antrum or body through endoscopic and pathological examinations, and multi-slice spiral CT scans revealed no distant metastasis. All case underwent totally laparoscopic distal gastrectomy with R anastomosis. Prospectively examined the intraoperative data, including operation time, time for R anastomosis, blood loss; Postoperative data including pathological data, duration of gastric tube placement, time to initiate liquid diet, the length of hospital stay; other functional outcomes and short-term postoperative complication data, graded according to the Clavien-Dindo complication classification system

ELIGIBILITY:
Inclusion Criteria:

(1) Elective surgery, indications for surgery: Cases diagnosed with malignant tumors of the gastric antrum or body by endoscopy and pathology, confirmed by multi-slice spiral CT to have no distant metastasis. (2) Patients who underwent laparoscopic distal gastrectomy with Billroth II + Braun anastomosis for gastric cancer, and can be followed up after surgery.

Exclusion Criteria:

(1) Patients who received neoadjuvant chemotherapy before surgery; (2) Emergency surgery patients; (3) Patients with concurrent malignant tumors; (4) Patients lost to follow-up due to non-tumor reasons after surgery.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases were confirmed to have malignant tumors in the gastric antrum or body through endoscopic and pathological examinations, and multi-slice spiral CT scans revealed no distant metastasis.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Complication | 6 months
  Anastomotic leakage;Anastomotic site bleeding;Anastomotic stenosis;Gastric emptying dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No